CLINICAL TRIAL: NCT06296238
Title: Nutrition and Inflammation in Pregnancy: Impacts on Early Human Brain Development in Ethiopia
Status: Completed | Type: Observational
Sponsor: Brown University (Other)
Collaborators: Addis Continental Institute of Public Health (Other); Boston Children's Hospital (Other); New York University (Other); Johns Hopkins University (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anne Shee CC Lee, Levinger Family Professor of Pediatrics, Brown University
Other Study IDs: 2023P000461
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Prenatal Exposure Delayed Effects
MeSH Terms: conditions — Prenatal Exposure Delayed Effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Enhanced Nutrition Package (ENP) health center + Enhanced Infection Management Package (EIMP): ENP: Health centers were strengthened to provide WHO/FMOH-recommended nutrition interventions in pregnancy. Pregnant women received a supply of adequately iodized salt for household use and iron-folate tablets from enrollment to birth. Women with undernutrition (MUAC <23 cm), also received a daily balanced energy protein supplement. EIMP: Pregnant women were screened at enrollment for bacteriuria with urine culture and antimicrobial susceptibility testing and presumptive deworming with mebendazole 500mg. Some women also received screening for chlamydia and gonorrhea and symptomatic women were tested for bacterial vaginosis and trichomonas. For women with chlamydia or gonorrhea, the participant was treated per FMOH guidelines with recommended antibiotics. STI/RTI screening was eventually discontinued due to supply shortage and the low prevalence of STI. At ANC follow-up visits, infected women were treated with antibiotics and persistent infection was retreated.
- ENP health center, routine care infection management participant: ENP: The health centers were strengthened to provide WHO/FMOH-recommended nutrition interventions in pregnancy. Pregnant women received a supply of adequately iodized salt for household use and iron-folate tablets from enrollment to birth. Women with undernutrition (MUAC <23 cm), also received a daily balanced energy protein supplement. Standard infection care: Maternal genitourinary tract infections is managed as per standard FMOH health center guidelines that utilize a syndromic management approach.
- Routine nutrition care health center, EIMP participant: Routine nutrition care: Maternal nutrition was managed as per standard FMOH health center guidelines.
  EIMP: Pregnant women were screened at enrollment for bacteriuria with urine culture and antimicrobial susceptibility testing and presumptive deworming with mebendazole 500mg. Some women also received screening for chlamydia and gonorrhea and symptomatic women were tested for bacterial vaginosis and trichomonas. For women with chlamydia or gonorrhea, the participant (and partner) was treated per FMOH guidelines with recommended antibiotics. STI/RTI screening was eventually discontinued due to supply shortage and the low prevalence of STI. At ANC follow-up visits, infected women were treated with antibiotics and persistent infection was retreated.
- Routine of care nutrition and infection management: Pregnant women received routine strengthened antenatal care services at the health center per FMOH guidelines. Maternal genitourinary tract infections were managed as per standard FMOH health center guidelines that utilize a syndromic management approach.

SUMMARY:
The goal of this observational child follow-up study is to examine the effects of prenatal nutrition and infection management interventions on long-term child neurodevelopment.

Participants are the offspring of mothers in the main study entitled "Enhancing Nutrition and Antenatal Infection Treatment (ENAT)" that was conducted in the rural Amhara region of Ethiopia. In the ENAT pragmatic clinical effectiveness study, 2399 pregnant women were randomized to receive routine prenatal care, a package of enhanced nutrition interventions (balanced energy protein supplement, iodized salt, iron-folic acid and counseling), a package of enhanced infection management interventions (genitourinary tract infection screening-treatment, deworming), or a combination of both packages. The impact of these antenatal nutrition and infection interventions on birth outcomes (infant birth size and gestational length) was examined in the main study. In this longitudinal cohort study, we will follow the offspring from the ENAT pregnancy cohort up to 24 months postnatal age and assess their growth, health and neurodevelopment.

The main questions it aims to answer are:

1. What are the effects of pregnancy interventions from the parent study (ENAT) on offspring neurodevelopmental outcomes?
2. What are the associations between maternal-newborn iron status and inflammation on infant neurodevelopment?
3. What are the associations between maternal iodine status and thyroid function on infant neurodevelopment?

We will follow children of mothers from the parent ENAT study to monitor their growth, health, and neurodevelopment up to 24 months postnatal age.

DETAILED DESCRIPTION:
In low-resource settings, undernutrition and infections during the first 1000 days of life are prevalent, modifiable risk factors that may have lifelong effects on a child's cognitive and psychological development, yet effective interventions addressing prevailing mechanisms are still to be validated. Iron, protein and energy are critical nutrients that support the rapidly developing fetal brain, however, among women of reproductive age in Sub-Saharan Africa, 10% are underweight and 20% have iron deficiency anemia. Pregnancy infections are also common in Africa, where one in three women have a geo-helminthic infection resulting in blood loss, iron deficiency and inflammation. The interaction between iron and inflammation in pregnancy is particularly complex. NICHD has identified the complex relationship between nutrition, inflammation, and neurodevelopment as a major research gap. A barrier to progress is that mechanistic understanding of prenatal brain development is based on animal or observational studies. We present a unique opportunity to leverage an ongoing randomized controlled trial (RCT) to examine the consequences of pregnancy nutrition and inflammation on child neurodevelopment.

The Enhancing Nutrition and Antenatal Infection Treatment (ENAT) RCT enrolled pregnant women in Amhara, Ethiopia to study independent and overlapping effects of prenatal nutrition and infection interventions on birth outcomes. Women were randomized to receive: 1) standard prenatal care, 2) enhanced nutrition package (ENP) (counseling, iron-folic acid [IFA], iodized salt, and balanced energy protein [BEP] supplementation), 3) enhanced infection management package (EIMP) (anti-helminthics, urinary tract infection treatment), or 4) ENP+EIMP. The current follow-up study (Longitudinal Infant Development and Growth; LIDG) will investigate biological pathways by which ENAT interventions, specifically iron, protein-energy, and inflammation, influence child neurodevelopment.

Our overarching hypotheses are that improving prenatal nutrition will improve brain structural and network development, reducing inflammation will improve white matter maturation, and the combination will have synergistic effects on child neuro-cognitive outcomes. This study will follow up to 500 ENAT children to assess neurodevelopment through 24 months of age, including neurobehavior and neural networks.

ELIGIBILITY:
Inclusion criteria:

* Mothers who have participated in ENAT study who consent to participate in the infant follow up study
* Intention to stay in the study catchment area
* Healthy infants without severe clinical signs or symptoms including headache, vomiting, or dizziness

Exclusion criteria:

* Major congenital anomalies
* Infants with severe morbidity or developmental disorder
* Neonatal encephalopathy
* Plan to move out of study catchment area

Ages: 9 Months to 27 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants of this study will be recruited from 6 rural health centers (serving a ~25,000 population) involved in ENAT study in West Gojjam and South Gondar zones, Amhara, Ethiopia (Lee et al., 2022). In this infant follow-up study, up to 500 selected infants from the parent ENAT study will be followed for 24 months for general health, growth, and development. A subset of these infants (up to 480) whose mothers provided biospecimens or whose mothers had mid-upper arm circumference (MUAC) of <23 cm in the parent study will be recruited for an advanced neurodevelopmental assessment study.
Sampling Method: Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Child resting brain function | 24 months
  Measured by absolute power of alpha frequency band on mobile electroencephalography

SECONDARY OUTCOMES:
Child resting brain function, secondary measures | 24 months
  Absolute and relative power of beta, theta, gamma frequency bands; relative alpha power, on mobile electroencephalography
Brain functional connectivity | 24 months
  Neural network efficiency and organization across brain regions measured by mobile electroencephalography
Neural processing speed | 24 months
  Visual Evoked Potential (VEP) P1 Latency
Visual Attention | 12 months
  Measured with infant eye tracking during Cecile Attention Task
Nonverbal Visual Attention | 12 months
  Multisensory Attention Assessment Protocol
Infant Neurologic Maturity | 12 months
  Hammersmith Infant Neurological Exam (HINE) Total Score
Infant Head Circumference | 12, 24 months
  Occipito-frontal head circumference
Child Cognitive Function | 24 months
  Bayley-III Cognitive Scale

CONTACTS AND LOCATIONS:
Overall Officials: Yemane Berhane, Principal Investigator — Addis Continental Institute of Public Health; Anne CC Lee, Principal Investigator — Warren Alpert Medical School of Brown University
Locations (1):
- Health Centers in West Gojjam and South Gondar zones, Bahir Dar, Amhara, Ethiopia

REFERENCES:
- [Derived] Roy Paladhi U, Workneh F, Baye E, Derebe MM, Yibeltal K, Fasil N, Driker S, Van Dyk F, I Chin T, North K, Jensen SKG, Christian P, Worku A, Berhane Y, Lee AC. Investigating biological mechanisms of adverse birth outcomes and early child development in Amhara, Ethiopia: protocol of biospecimen collection and analysis of the Enhancing Nutrition and Antenatal Infection Treatment (ENAT) randomised effectiveness study. BMJ Open. 2025 Apr 28;15(4):e098686. doi: 10.1136/bmjopen-2024-098686. PMID 40295129
- [Derived] Workneh F, Chin TI, Yibeltal K, Fasil N, North K, Jensen SKG, Kidane WT, Melese M, Tsegaye S, Berhane YY, Roy Paladhi U, Abate BH, Teklehaimanot A, Melka TL, Pihl S, An WW, Van Dyk F, Mullany LC, Folger LV, Cherkerzian S, Troller-Renfree SV, Thomason ME, Andersson M, Inder T, Nelson CA, Grant PE, Christian P, Worku A, Berhane Y, Lee AC. Impact of maternal antenatal nutrition and infection treatment interventions on Longitudinal Infant Development and Growth in rural Ethiopia: protocol of the LIDG child follow-up study. BMJ Paediatr Open. 2024 Dec 24;8(1):e002840. doi: 10.1136/bmjpo-2024-002840. PMID 39725450